CLINICAL TRIAL: NCT04514432
Title: Mindful Melody: Feasibility of Implementing Music Listening on an Inpatient Psychiatric Unit and Its Relation to the Use of As Needed Medications for Acute Agitation
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Luba Leontieva, Assisstant Professor of Psychiatry, State University of New York - Upstate Medical University
Other Study IDs: 1434789-1
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Agitated; State, Acute Reaction to Stress; Agitation,Psychomotor
Keywords: Agitation; Music; Inpatient
MeSH Terms: conditions — Psychomotor Agitation; Stress Disorders, Traumatic, Acute | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- When music was available: 3 month period during which music was available to patients experiencing agitation
  Interventions: Other: Music
- When music was not available: 3 month period during which music was not available to patients

INTERVENTIONS:
Other: Music — If patients experienced agitation, they were able to request to listen to music for 30 minutes. They listened to genre playlists generated by the music application Spotify.
  Groups: When music was available

SUMMARY:
In this quality improvement project, our objectives were to assess the feasibility and effectiveness of using music as an adjunct to or replacement of pharmacological interventions for patient agitation on an inpatient psychiatric unit. We hypothesized that music availability would help to reduce agitation and reduce the amount of as-needed medications used for cases of patient agitation.

DETAILED DESCRIPTION:
The number of as-needed medications for agitation was quantified during a three month period during which patients had the option of listening to music in cases of agitation. This was compared to the number of medications needed for agitation during another 3 month period during which music was not available. The medications used were quantified using pharmacy records. Patients and nurses were surveyed to determine how effective and feasible they thought the music intervention was. The study was conducted at the SUNY Upstate University Hospital inpatient psychiatric unit, which is a 24-bed unit. 172 patients were included in the project.

Before starting to offer music, a basic training meeting was held with nursing staff to understand the purpose of the project. Patients participating had the option of selecting a preferred musical genre and they listened to music using wireless headphones. The playlists used were genre playlists automatically generated by Spotify music application. If patients did not like the song that was generated, they had an option to skip the song using their bluetooth headphone controls. Headphones were collected after 30 minutes of listening unless they were return prior to completion of the listening session.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 18 years or older admitted to the inpatient psychiatric unit

Exclusion Criteria:

* Patients who did not want to listen to music or be included in the project were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: inpatients on an acute psychiatric unit
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
The number of medications used for agitation | 5/18/2018 until 11/13/2018
  The number of different types of medications used for agitation was quantified using pharmacy records

SECONDARY OUTCOMES:
Scales administered to nursing staff | 5/18/2018 until 11/13/2018
  Scales administered to nursing to determine ease of implementation and effect on the psychiatric unit milieu
Scales administered to patients | 5/18/2018 until 11/13/2018
  Scales administered to patients to assess the extent of the calming effect of listening to music

CONTACTS AND LOCATIONS:
Locations (1):
- Upstate University Hospital, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scudamore T, Liem A, Wiener M, Ekure NS, Botash C, Empey D, Leontieva L. Mindful Melody: feasibility of implementing music listening on an inpatient psychiatric unit and its relation to the use of as needed medications for acute agitation. BMC Psychiatry. 2021 Mar 6;21(1):132. doi: 10.1186/s12888-021-03127-z. PMID 33676455